CLINICAL TRIAL: NCT05399797
Title: Impact of Online Counselling Training For Pharmacists on The Management of Acute Uncomplicated Urinary Tract Infections in Adults; A Double-blind Randomized Controlled Trial
Brief Title: Management of Acute Uncomplicated UTIs in Adults by Community Pharmacists
Acronym: [UTI]
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Ibadan (Other)
Responsible Party: Principal Investigator, Abdulhafiz Taofiq Tanimola, Principal Investigator, University of Ibadan
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Health Services Research
Other Study IDs: taofiqclinical
Record Dates: First submitted 2022-05-07; First posted 2022-06-01 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Urinary Tract Infections; Urinary Tract Infection Lower Acute
Keywords: Urinary Tract Infections; Pharmacist; Mystery Patient
MeSH Terms: conditions — Urinary Tract Infections | interventions — Training Support

STUDY DESIGN:
Intervention Model Description: The pharmacists in the interventional group will receive educational training after baseline assessment while those in the control group will receive the same training at the end of the study
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The participating pharmacists, the mystery patient and the investigator will not know who is in the control or the intervention group
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pharmacists in the intervention group (Experimental): The pharmacist will be given an online educational training on management of acute uncomplicated urinary tract infections
  Interventions: Other: Educational training
- Pharmacists in the control group (No Intervention): pharmacists in this group will not be trained, until after the completion of the study.

INTERVENTIONS:
Other: Educational training — Pharmacists in the intervention group will given detailed online educational training on how to recognize and manage acute uncomplicated urinary tract infections in adults.
  Arms: Pharmacists in the intervention group

SUMMARY:
This study is to be conducted in community pharmacies. It involves the use of trained mystery patients to evaluate community pharmacists at baseline and post intervention. The pharmacists will be divided into control and intervention groups using computer generated codes. Those in the intervention group will receive an online training by clinical pharmacists. The training will employ the use of didactic teaching and the use of case studies and simulations covering the diagnosis and management of acute uncomplicated urinary tract infections in adults. Post intervention, mystery patients will revisit the community pharmacists in the control and intervention groups for re-assessment.

ELIGIBILITY:
Inclusion Criteria:

* The superintendent pharmacist, or the pharmacist manager or any other post National Youth Service Corps pharmacist

Exclusion Criteria:

* Interns, and pharmacists undergoing the mandatory National Youth Service Corps program.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2022-03-21 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2022-11 (Estimated)

PRIMARY OUTCOMES:
Questioning skill score | Through the study completion (an average of 6 months)
  Expert Panels' Relevant Questions - Through 80% consensus the expert panel picked 50 relevant questions. The minimum score is "0" and the maximum score is "50". The higher the score the better the questioning skill.
Correct diagnosis of Acute Uncomplicated Urinary Tract Infection | Through the study completion (an average of 6 months)
  using the Infectious Disease Society of America treatment guideline, the pharmacists should be able to reach a diagnosis of Acute Uncomplicated Urinary Tract Infection. Appropriate diagnosis will be classified as "Correct diagnosis" and inappropriate diagnosis will be classified as "Incorrect diagnosis". Proportion will be used to describe the number of community pharmacists who got the diagnosis Correct and Incorrect.
Appropriate management of urinary tract infection | Through the study completion (an average of 6 months)
  Infectious Disease Society of America treatment guideline

CONTACTS AND LOCATIONS:
Overall Officials: Segun J Showande, Ph.D., Study Chair — University of Ibadan
Locations (1):
- University of Ibadan, Ibadan, Oyo State, Nigeria

IPD SHARING:
Plan to Share IPD: No